CLINICAL TRIAL: NCT00770107
Title: Thiamine Supplementation to Improve Cardiac Function in Patients With Congestive Heart Failure on Long-term Treatment With Diuretic Drugs
Brief Title: Thiamine Supplementation to Improve Cardiac Function in Patients With Congestive Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Paul Erne, Kantonsspital Luzern
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Thiamine in Heart Failure
Record Dates: First submitted 2008-10-03; First posted 2008-10-09 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Thiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Thiamine (Active Comparator)
  Interventions: Drug: Thiamine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thiamine — Supplementation of thiamine (vitamin b1) 300 mg per day, once daily, for a duration of 4 weeks
  Arms: Thiamine
Drug: Placebo — Placebo, once daily, for a duration of 4 weeks
  Arms: Placebo

SUMMARY:
Working Hypothesis: a treatment with thiamine improves functional status and heart function of patients with congestive heart failure when on a diuretic treatment.

DETAILED DESCRIPTION:
In the treatment of congestive heart failure, diuretic drugs have become a firm cornerstone of therapy. Up to 50% of patients with congestive heart failure in industrialized nations will undergo long-term diuretic treatment. Diuretic therapy is associated with a loss of water soluble vitamins, including vitamin B1 (thiamine). Electrolyte dysbalance, a major side effect of diuretic therapy, has been extensively studied. In sharp contrast, only few data are available about the effects of vitamin loss and in particular of thiamine in this setting. Available data suggest that a diuretic treatment is associated with an increased risk for thiamine deficiency. Thiamine plays a crucial role for normal cardiac function, since severe thiamine deficiency leads to congestive heart failure (wet beriberi). Consequently, patients undergoing diuretic treatment might have compromised heart function. Supplementation of thiamine has been reported to improve cardiac function in patients with congestive heart failure on long-term treatment with diuretic drugs. However, no efforts have been made to confirm those preliminary observations by a placebo-controlled, double-blind study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable congestive heart failure on a prescription for diuretic drugs

Exclusion Criteria:

* Acute heart failure
* Foreseeable need for further changes in medication
* Current medication containing vitamins
* Patients with a creatinine above 250 μmol/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2004-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | One day, one week, two weeks, four weeks

SECONDARY OUTCOMES:
Quality of life | One day, one week, two week, four weeks
6-minutes walking test | One day, one week, two weeks, four weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Luzern, Lucerne, Canton of Lucerne, Switzerland

REFERENCES:
- [Derived] Schoenenberger AW, Schoenenberger-Berzins R, der Maur CA, Suter PM, Vergopoulos A, Erne P. Thiamine supplementation in symptomatic chronic heart failure: a randomized, double-blind, placebo-controlled, cross-over pilot study. Clin Res Cardiol. 2012 Mar;101(3):159-64. doi: 10.1007/s00392-011-0376-2. Epub 2011 Nov 5. PMID 22057652